CLINICAL TRIAL: NCT04074681
Title: Efficacy of an Internet-based Psychological Intervention for Problem Gambling and Gambling Disorder: A Randomized Controlled Trial
Brief Title: Efficacy of an Internet-based Psychological Intervention for Problem Gambling and Gambling Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UJI-A2016-14
Record Dates: First submitted 2019-07-22; First posted 2019-08-30 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Pathological Gambling
Keywords: Gambling; CBT; Internet program; Efficacy
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gambling Internet-based Protocol (Experimental): Intervention group that carries out the Gambling Internet-based Protocol based on Cognitive and Behavioral Therapy (CBT) and receives support by the therapist (a weekly 10-minute phone call without clinical content). In addition, they will receive one notification per day to respond to the EMI questions at 8 PM. The EMI includes immediate automatic feedback depending on the participant's responses.
  Interventions: Behavioral: Gambling Internet-based Protocol
- Waiting List Control Group (No Intervention): Participants in a 12-week waiting list control condition. They will be offered the possibility of receiving the online treatment protocol after the waiting list period.

INTERVENTIONS:
Behavioral: Gambling Internet-based Protocol — Gambling Internet-based protocol is a multimedia interactive and self-help program for problem and pathological gamblers, which will allow individuals to learn and practice adaptive ways to cope with this problem. The main therapeutic modules included in this program are: 1) Motivational for change; 2) Psychoeducation; 3) Stimulus control (e.g. self-prohibition and blocking of usual gambling websites with therapist confirmation) and responsible return of debts; 4) Cognitive restructuring; 5) Emotion regulation; 6) Planning of significant activities; 7) Coping skills and exposure with response prevention; 8) Relapse prevention.
  Arms: Gambling Internet-based Protocol

SUMMARY:
The aim of this study is to assess the efficacy of an online CBT-based intervention combined with an Ecological Momentary Intervention (EMI) and different complementary tools for the treatment of problem gambling and gambling disorder. The main hypothesis is that the Internet-based psychological intervention group will obtain better results than the waiting list control group.

DETAILED DESCRIPTION:
Gambling Disorder is a prevalent non-substance use disorder, which contrasts with the low number of people requesting treatment. Information and Communication Technologies (ICT) could help to enhance the dissemination of evidence-based treatments and considerably reduce the costs. The current study seeks to assess the efficacy of an online psychological intervention for people suffering from gambling problems in Spain. The proposed study will be a two-arm, parallel-group, randomized controlled trial. A total of 134 participants (problem and pathological gamblers) will be randomly allocated to a waiting list control group (N=67) or an intervention group (N=67). The intervention program includes 8 modules, and it is based on motivational interviewing, cognitive-behavioural therapy (CBT), and extensions and innovations of CBT. It includes several complementary tools that are present throughout the entire intervention. Therapeutic support will be provided once a week through a phone call with a maximum length of 10 minutes. The primary outcome measure will be gambling severity and gambling-related cognitions, and secondary outcome measures will be readiness to change, and gambling self-efficacy. Other variables that will be considered are depression and anxiety symptoms, positive and negative affect, difficulties in emotion regulation strategies, impulsivity, and quality of life. Individuals will be assessed at baseline, post-treatment, and 3-, 6-, and 12-month follow-ups. During the treatment, participants will also respond to a daily Ecological Momentary Intervention (EMI) in order to evaluate urges to gamble, self-efficacy to cope with gambling urges, gambling urge frequency, and whether gambling behaviour occurs. The EMI includes immediate automatic feedback depending on the participant's responses. Treatment acceptance and satisfaction will also be assessed. The data will be analysed both per protocol and by Intention-to-treat. As far as we know, this is the first randomized controlled trial of an online psychological intervention for gambling disorder in Spain. It will expand our knowledge about treatments delivered via the Internet and contribute to improving treatment dissemination, reaching people suffering from this problem who otherwise would not receive help.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older.
* Willingness to participate in the study and sign informed consent.
* To have and handle the computer, Internet and an email address.
* Ability to understand, read and write Spanish.
* Based on the cut-off points established by the Norc diagnostic screen for gambling disorders (NODS; adapted by Becoña, 2004): be a problem gambler (3-4 items) or a pathological gambler (5 or more items).
* Willingness to provide the name of a co-therapist to validate the information provided, as well as to be able to locate the patient in follow-ups.
* Willing to provide follow-up data on gambling.

Exclusion Criteria:

* Any serious mental disorder (Bipolar and Related Disorders and Schizophrenia Spectrum and Other Psychotic Disorders), medical illness, and moderate or severe alcohol and/or substance use disorder, that prevents the program from being carried out.
* If their gambling behaviour occurs in the context of a Maniac Episode or because of the intake of dopaminergic medication (e.g. Parkinson's disease).
* The presence of high suicidal risk.
* Receiving another psychological treatment while the study is still ongoing.
* Receiving pharmacological treatment is not an exclusion criterion during the study period, but participants having an increase and/or change in the medication 2 months prior to enrollment will not be considered for the trial. Also, the increase and/or change in the medication during the study period in the experimental group will imply the participant's exclusion from subsequent analyses (a decrease in pharmacological treatment is accepted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Gambling Symptom Assessment Scale (G-SAS; Kim, Grant, Potenza, Blanco & Hollander, 2009) at Pre-intervention, Post-module, Post-intervention, 3-, 6-, and 12 months Follow-up. | Up to 12 months
  The G-SAS is a 12-item self-report instrument that assesses gambling symptom severity. All items are referred to as an average symptom based on the past 7 days.The statements correspond with gambling urges;average frequency, duration,and control of thoughts associated with gambling;time spent on gambling or gambling-related behaviour;anticipatory excitement caused by an imminent gambling act; pleasure associated with winning;emotional distress;and personal trouble.All items are rated on a 4-point scale (total score: 0-48).The higher score the higher gambling symptoms severity (mild=8-20;moderate=21-30;severe=31-40;extreme=41-48).It shows high internal consistency (α=0.87) and good convergent validity with other measures associated with gambling symptom severity in a sample of pathological gamblers.Because this instrument has not a Spanish version, standardized procedures were followed to adapt G-SAS to the Spanish language.Cronbach's alpha will be calculated with the data at hand.
Change in the Gambling-Related Cognitions Scale (GRCS-S; Raylu & Oei, 2004; Spanish validation Del Prete, Steward, Navas, Fernández-Aranda, Jiménez-Murcia, Oei & Perales, 2016) at Pre-intervention, Post-intervention, 3-, 6-, and 12 months Follow-up. | Up to 12 months
  The GRCS-S is a self-report instrument aimed to assess five domains of gambling-related cognitions (interpretative bias, IB; the illusion of control, IC; predictive control, PC; gambling expectancies, GE; and perceived inability to stop gambling, ISG). It comprises 23 items which are worded on a 7-point Likert type scale (1= I completely disagree; 7=I completely agree). The total score consists of adding the values of the whole items. The score for each subscale is obtained adding the values for the items' set that represent each subscale. The higher the total score the higher the number of gambling-related cognitions presented. GRCS-S shows adequate psychometric properties in a sample composed by treatment-seeking gamblers and non-treatment-seeking gamblers: the concurrent and criterion-related validity are verified, the full scale reliability is 0.95, and for each subscale reliability ranges from 0.68 to 0.91 (GE= 0.77; IC=0.68; PC=0.84; ISG=0.91; IB= 0.89).

SECONDARY OUTCOMES:
Change in the Gambling Self-Efficacy Questionnaire (GSEQ; May, Whelan, Steenbergh & Meyers, 2003; Winfree, Ginley, Whelan, & Meyers, 2014) at Pre-intervention, Post-module, Post-intervention, 3-, 6-, and 12 months Follow-up. | Up to 12 months
  The GSEQ is a self-report instrument that assesses perceived self-efficacy to control gambling in high-risk situations through 16 six-point Likert scale items. Participants are asked to indicate how confident they feel in a scale that ranges from 0% (Not at all confident) to 100% (Very confident) in increments of 20%. Specifically, it includes intrapersonal (e.g. unpleasant emotions, physical discomfort, pleasant emotions, testing personal control, and urges and temptations) and interpersonal factors (conflict with others, social pressure and pleasant times with others) based on Marlatt's (1985) model of relapse situations for addictive behaviors. The overall score is calculated taking into account the mean response from all items, and it can range from 0 to 100. The higher overall score the higher overall confidence about controlling their gambling behavior. There is evidence of convergent and discriminant validity, and the internal consistency is high (α=0.99) in a community sample.
Change in the University of Rhode Island Change Assessment Scale (URICA; McConnaughy, Prochaska & Velicer, 1983; Spanish validation Gómez-Peña et al., 2011) at Pre-intervention, Post-intervention, 3-, 6-, and 12 months Follow-up. | Up to 12 months
  The URICA is a 32 items self-report instrument that includes four subscales and assesses four of the five stages of change proposed by Prochaska & DiClemente (precontemplation, PC; contemplation, C; action, A; and maintenance, M) on a 5-point Likert type scale (1=strongly disagree; 5=strongly agree). Scores for each subscale range from 8 to 40, and are obtained adding the value of the 5 items that include each subscale. A second-order score is obtained and is referred to the degree of 'Readiness to change' (C+A+M-PC). The URICA shows good psychometric proprieties in a sample of pathological gamblers. The internal consistency values are adequate for the stages of change assessed as well as for the total score corresponding to 'Readiness to change'. Specifically, the Cronbach's alpha coefficients ranges from 0.74 to 0.84 taking into account the different stages (Precontemplation=0.74; Contemplation=0.80; Action=0.84; and Maintenance=0.74) and for the total score is 0.84.
Change in the EMI measures during procedure. | During procedure.
  Gambling urge intensity (on a scale from 0 "Not at all" to 10 "maximum") and frequency (on a 5-point Likert scale from "Never" to "Almost always"), self-efficacy to cope with gambling urges (on a scale from 0 "Not at all" to 10 "Completely"), gambling behaviour (yes/no), money wagered (euros), and amount of time gambling (minutes) are also assessed for 90 days in the experimental group.

OTHER OUTCOMES:
Change in the NORC DSM-IV Screen for Gambling Problems (NODS; Gernstein et al., 1999; Becoña, 2004) at Pre-intervention (screening), Post-intervention, 3-, 6- and 12 months Follow-up. | Up to 12 months
  The NODS is a hierarchically structured 17-item screen that is designed to assess the at-risk, problem and pathological gambling. It is referred to the experience in gambling both throughout their life and in the last year, with dichotomous choice questions (Yes / No). The total score ranges from 0 to 10 (1-2 affirmative items correspond with at-risk gambling; 3-4 items with problem gambling; and 6 or more with pathological gambling). The data obtained on specificity and sensitivity is good, its test-retest reliability is 0.98, and its validity is excellent considering that it corresponds strictly to the DSM-IV criteria. We will use the 12-month version at pre-test to establish the diagnosis based on the DSM-IV-TR, and the 3-month version of the NODS to assess the progress made in gambling severity throughout the intervention and in follow-up assessments.
Mini International Neuropsychiatric Interview - The M.I.N.I. 7.0.2, 8/8/16 version (Sheehan, 2016). | Pre-intervention (screening)
  MINI is a brief structured diagnostic interview and is designed to assess the most common psychiatric disorders in ICD-10 and DSM-5 (major depressive episode; obsessive-compulsive disorder; posttraumatic stress disorder; alcohol use disorder; substance use disorder; any psychotic disorder; anorexia nervosa; bulimia nervosa; generalized anxiety disorder; medical, organic, drug cause ruled out; and antisocial personality disorder). Questions are rated dichotomously (yes/no) and clinical judgment should be used in coding the responses, asking for examples if it is needed. Validity and reliability are supported and similar properties to the SCID-P for DSM-III-R and the CIDI are shown, but it can be administered in a much shorter period of time.
Gambling history interview and current gambling situation and related variables assessment at the pre-intervention (screening) | Pre-intervention (screening)
  This interview is based on the Structured Interview of Gambling History (Echeburúa & Báez, 1994). In addition to making a selection of five of the items of the first interview to assess parents' gambling habits, the onset, and aggravation of the patient's gambling behaviour (including ups and downs and periods of abstinence), other five interesting items of variables related to the current gambling situation are added. They are referred to economic debts, to which people or entities they owe money and the specific amount, if they have access to money and the forms through which they can access, what they have done so far to solve the problem, how long it has happened since the last bet and the specific risk places. The 10 items are open-ended questions and offer qualitative data to understand the participants' context and gambling situation.
Change in the Hospital Anxiety Depression Scale (HADS) (Zigmond and Snaith, 1983; Castresana et al., 1995) at Pre-intervention, Post-intervention, 3-, 6-, and 12 months Follow-up. | Up to 12 months
  HADS is a self-report instrument that consists of 14 items and has two subscales: seven items measure depressive symptoms and the other seven items anxiety symptoms. Respondents are asked to indicate which option fits them the most, taking the past week into account. Each item is rated in a four-point scale from 0 to 3. The scores for both subscales are obtained by adding all the items values, and both ranges from 0 to 21. Scores up to 8 indicates there is absence of significant morbidity, from 8 to 10 corresponds to a borderline case, and scores higher than 10 indicates morbidity. The internal consistency rates from 0.42 to 0.71 (p<0.01) regarding depression subscale, and from 0.36 to 0.64 regarding anxiety subscale.
Change in the Overall Depression Severity and Impairment Scale (ODSIS; Bentley, Gallagher, Carl & Barlow, 2014; Spanish validation Mira et al., 2019) at Post-module. | During procedure.
  ODSIS is a 5-item self-report instrument that evaluates a unidimensional factor referred to the severity and functional impairment associated with depression during the last week. There are five response options for each item and they are coded from 0 to 4. The total score is obtained adding the values of all the items and it ranges from 0 to 20. Scores of 5 or higher indicate depressive symptoms. This scale is validated online considering a sample of patients with depressive or anxiety disorders. It shows an excellent internal consistency (α=0.92), and the construct, convergent and discriminant validities are evidenced.
Change in the Overall Anxiety Severity and Impairment Scale (OASIS; Campbell-Sills et al., 2009; Spanish validation González-Robles et al., 2018) at Post-module. | During procedure.
  OASIS is a 5-items self-report instrument that assesses a unidimensional factor referred to the severity and frequency of anxiety symptoms, as well as to the behavioral avoidance and the functional impairment related to these symptoms in the previous week. There are five response options for each item and they are coded from 0 to 4. The total score is obtained adding the values of all the items and it ranges from 0 to 20. Scores higher than 8 show the occurrence of anxiety symptoms. This scale is validated online in a sample of patients with depression and anxiety. It shows good internal consistency (α=0.86) and adequate convergent and discriminant validities, as well as sensitivity to change.
Change in the Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004: Spanish validation Hervás & Jódar, 2008) at Pre-intervention, Post-intervention, 3-, 6-, and 12 months Follow-up. | Up to 12 months
  DERS is a self-report measure that includes 28 items and it assesses five factors related to difficulties in emotion regulation processes: emotional lack of control, life interference, lack of emotional attention, emotional confusion, and emotional rejection. Participants should report in a 5-point Likert type scale how often the items are applied for themselves from 1 (almost never; 0-10%) to 5 (almost always; 91-100%). A score for each subscale is obtained adding the values of the set of items that correspond to each subscale and taking into account reversed items. A final score is obtained adding the values of all items. The higher scores the higher difficulties in emotion regulation processes. DERS has good psychometric properties in the general population. Internal consistency is 0.93, test-retest reliability is adequate, and convergent and incremental validities are evidenced.
Change in the Positive and Negative Affect Schedule (PANAS; Watson, Clark & Tellegen, 1988) at Pre-intervention, Post-intervention, 3-, 6-, and 12 months Follow-up. | Up to 12 months
  The PANAS is made up of 20 items that assess two independent dimensions, positive affect (PA) and negative affect (NA). PANAS is used for measuring trait and state affectivity. Each dimension consists of 10 items which are rated on a 5-point Likert type scale (1=very slightly or not at all; 2= a little; 3=moderately; 4; quite a bit; 5=very much). Participants should indicate to what extent they have experienced each emotion generally and during the last week. Total scores are calculated adding the values of the items for each dimension, and it ranges from 10 to 50. Psychometric properties are not yet available since the Spanish validation in clinical patients is ongoing, but Cronbach's alpha will be calculated with the data at hand.
Change in the Short UPPS-P Impulsivity Scale (UPPS-P; Lynam, Smith, Whiteside & Cyders, 2006; Spanish validation Cándido, Orduña, Perales, Verdejo-García & Billieux, 2012) at Pre-intervention, Post-intervention, 3-, 6-, and 12 months Follow-up. | Up to 12 months
  UPPS-P assess five impulsivity traits (negative urgency, lack of premeditation, lack of perseverance, sensation seeking and positive urgency) through 20 four-point Likert scale items (1=strongly agree; 4=strongly disagree). Scores of each of the five factors and a global score of the UPPS-P are obtained taking into account direct and inverse items. It is calculated adding the values of the four items that include each factor. The higher the score the higher impulsivity. UPPS-P present good psychometric properties in a sample of university students. Internal consistency is acceptable (α ranges from 0.61 to 0.81) and external validity is supported.
Change in the Quality Life Index (QLI; Mezzich, Cohen & Ruipérez, 1999; Spanish validation Mezzich, Ruipérez, Pérez, Yoon, Liu & Mahmud, 2000) at Pre-intervention, Post-intervention, 3- , 6-, and 12 months Follow-up. | Up to 12 months
  QLI is a 10-item self-report instrument that assess one concept of quality of life taking into account 10 dimensions on a ten-point Likert type scale (1=poor; 10=excellent): physical well-being, psychological/emotional well-being, self-care and independent functioning, occupational functioning, interpersonal functioning, social-emotional support, community and services support, personal fulfillment, spiritual fulfillment and global perception of quality of life. Total score corresponds to the average of the scores of the set of items and rages from 1 to 10 (1-4,5=perception of the quality of life below the average; 4,6-8,1= perception of the quality of life in the average; 8,2-10=perception of the quality of life above average). Internal consistency (α=0.89) and test-retest reliability (0.89) are high, and the discriminant validity is evidenced in a sample of psychiatric patients.
Change in the System Usability Scale (SUS; Castilla et al., 2016) after the first use of the program (after the welcome module) and post-intervention. | Up to 3 months
  SUS is a 10-item self-report instrument aimed to assess the system usability opinion in a 5-Likert type scale that ranges from 1 ( Completely disagree) to 5 (Completely agree). Psychometric properties are not yet available since the Spanish validation in clinical patients is ongoing, but Cronbach's alpha will be calculated with the data at hand.

CONTACTS AND LOCATIONS:
Overall Officials: Juana M Bretón López, Lecturer, Study Director — Universitat Jaume I; Azucena García Palacios, Lecturer, Study Director — Universitat Jaume I

REFERENCES:
- [Background] Bucker L, Bierbrodt J, Hand I, Wittekind C, Moritz S. Correction: Effects of a depression-focused internet intervention in slot machine gamblers: A randomized controlled trial. PLoS One. 2018 Aug 23;13(8):e0203145. doi: 10.1371/journal.pone.0203145. eCollection 2018. PMID 30138469
- [Background] Carlbring P, Smit F. Randomized trial of internet-delivered self-help with telephone support for pathological gamblers. J Consult Clin Psychol. 2008 Dec;76(6):1090-4. doi: 10.1037/a0013603. PMID 19045977
- [Background] Hodgins DC, Cunningham JA, Murray R, Hagopian S. Online Self-Directed Interventions for Gambling Disorder: Randomized Controlled Trial. J Gambl Stud. 2019 Jun;35(2):635-651. doi: 10.1007/s10899-019-09830-7. PMID 30701377
- [Background] Goslar M, Leibetseder M, Muench HM, Hofmann SG, Laireiter AR. Efficacy of face-to-face versus self-guided treatments for disordered gambling: A meta-analysis. J Behav Addict. 2017 Jun 1;6(2):142-162. doi: 10.1556/2006.6.2017.034. PMID 28662618
- [Derived] Diaz-Sanahuja L, Campos D, Mira A, Castilla D, Garcia-Palacios A, Breton-Lopez JM. Efficacy of an internet-based psychological intervention for problem gambling and gambling disorder: Study protocol for a randomized controlled trial. Internet Interv. 2021 Oct 5;26:100466. doi: 10.1016/j.invent.2021.100466. eCollection 2021 Dec. PMID 34646753
- See also: Laboratory of Psychology and Technology of the Jaume I University — http://www.labpsitec.uji.es